### over letter

### tle of the study

re the results of patient reported outcome measures after spine surgery influenced by recall of preoperative scores? – andomized controlled trial

**)** :HSJ1989

### late of the document

February 1, 2021

### Sample size calculation

- Primary endpoint: postoperative COMI
- Secondary endpoints: postoperative ODI/NDI and EQ5D
- Objective: compare means of PROMs between two groups according to the presence of recall of postoperative status in questionnaires
- Sample size was calculated for two sided T-test sig. level of 0.05, power of 0.80
- Effect size calculated according to Cohen's d = (M2 M1)/SD. The MCID for COMI (pt) is 1.7 = (M2 M1) (https://doi.org/10.1007/s00586-011-2100-3). We based the SD (2.7-2.9) for postoperative COMI in patients with lumbar surgeries in this work: https://doi.org/10.1007/s00586-018-5469-4.
- d = 1.7/2.8 = 0.61
- The calculated sample size was 86 patients (43\*2).

```
wr.t.test(d = 0.61, sig.level = 0.05, power = 0.8, type = "two.sample
")

Two-sample t test power calculation

n = 43.16853
d = 0.61
sig.level = 0.05
power = 0.8
alternative = two.sided

NOTE: n is number in *each* group
```

# Patient characteristics by group (overall = cervical+lumbar)

- Groups: Postoperative questionnaires; Postoperative questionnaires with recall of preoperative patient answers
- The groups have the same baseline characteristics, except for age but without clinical significance (57 y vs 60 y)
- Patients without recall report worse postoperative scores for COMI, ODI/NDI and EQ5D
- However this did not happened for mean of improvement for each score
- Also, the groups had the same perceived outcomes by the patients and similar satisfaction grades (outcomes perceived by the patient are slight better in recall group, but with no statistic significance)

| | no recall (N=75) | recall (N=74) |
|---|---|---|
| Gender | | |
| Female | 43 (57.3%) | 46 (62.2%) |
| Male | 32 (42.7%) | 28 (37.8%) |
| Age | | |
| Mean (SD) | 56.987 (10.112) | 60.527 (11.408) |
| Median (Q1, Q3) | 56.000 (49.000, 63.000) | 62.000 (52.250, 69.000) |
| Pathology | | |
| myelopathy | 25 (33.3%) | 20 (27.0%) |
| myelopathy/radiculopathy | 8 (10.7%) | 6 (8.1%) |
| neurogenic claudication | 7 (9.3%) | 14 (18.9%) |
| radiculopathy | 5 (6.7%) | 4 (5.4%) |
| sciatic pain | 24 (32.0%) | 23 (31.1%) |
| sciatic pain/neurogenic claudication | 6 (8.0%) | 7 (9.5%) |
| ВМІ | | |
| Mean (SD) | 27.511 (4.053) | 27.711 (4.411) |
| Median (Q1, Q3) | 27.275 (25.325, 29.888) | 26.930 (24.800, 29.670) |
| Smoker | | |
| yes | 15 (20.3%) | 9 (12.5%) |
| no | 59 (79.7%) | 63 (87.5%) |
| gment | | |

| | no recall (N=75) | recall (N=74) |
|----------------------|-------------------------|-------------------------|
| Cervical | 38 (50.7%) | 30 (40.5%) |
| Lumbar | 37 (49.3%) | 44 (59.5%) |
| Segment and group | | |
| Cervical no recall | 38 (50.7%) | 0 (0.0%) |
| Cervical with recall | 0 (0.0%) | 30 (40.5%) |
| Lumbar no recall | 37 (49.3%) | 0 (0.0%) |
| Lumbar with recall | 0 (0.0%) | 44 (59.5%) |
| preop COMI | | |
| Mean (SD) | 7.735 (1.859) | 7.512 (1.874) |
| Median (Q1, Q3) | 8.000 (6.500, 9.000) | 8.000 (7.000, 9.000) |
| preop ODI/NDI | | |
| Mean (SD) | 51.837 (19.223) | 47.068 (17.539) |
| Median (Q1, Q3) | 53.000 (40.000, 64.200) | 48.000 (37.780, 58.000) |
| preop EQ5D | | |
| Mean (SD) | 0.339 (0.336) | 0.399 (0.306) |
| Median (Q1, Q3) | 0.516 (-0.010, 0.587) | 0.516 (0.089, 0.620) |
| postop COMI | | |
| Mean (SD) | 5.479 (2.678) | 4.406 (2.778) |

| | no recall (N=75) | recall (N=74) |
|----------------------|-------------------------|-------------------------|
| Median (Q1, Q3) | 5.000 (4.000, 8.000) | 4.000 (2.000, 6.000) |
| postop ODI/NDI | | |
| Mean (SD) | 37.995 (20.314) | 29.023 (19.029) |
| Median (Q1, Q3) | 36.000 (22.500, 53.825) | 28.000 (14.000, 39.000) |
| postop EQ5D | | |
| Mean (SD) | 0.503 (0.314) | 0.609 (0.325) |
| Median (Q1, Q3) | 0.587 (0.516, 0.691) | 0.689 (0.516, 0.812) |
| Education | | |
| <=4 | 26 (48.1%) | 24 (47.1%) |
| >4 | 28 (51.9%) | 27 (52.9%) |
| Satisfaction.numeric | | |
| Mean (SD) | 4.528 (1.074) | 4.493 (1.146) |
| Median (Q1, Q3) | 5.000 (5.000, 5.000) | 5.000 (5.000, 5.000) |
| Outcome.numeric | | |
| Mean (SD) | 3.694 (1.182) | 3.986 (1.050) |
| Median (Q1, Q3) | 4.000 (3.000, 5.000) | 4.000 (3.000, 5.000) |
| Odom.numeric | | |
| Mean (SD) | 2.560 (0.904) | 2.635 (0.930) |

| | no recall (N=75) | recall (N=74) |
|---|---|---|
| Median (Q1, Q3) | 3.000 (2.000, 3.000) | 3.000 (2.000, 3.000) |
| Satisfaction | | |
| N-Miss | 3 | 5 |
| very dissatisfied | 4 (5.6%) | 4 (5.8%) |
| somewhat dissatisfied | 2 (2.8%) | 3 (4.3%) |
| neither satisfied or dissatisfied | 2 (2.8%) | 3 (4.3%) |
| somewhat satisfied | 8 (11.1%) | 4 (5.8%) |
| very satisfied | 56 (77.8%) | 55 (79.7%) |
| Outcome | | |
| N-Miss | 3 | 5 |
| made things worse | 5 (6.9%) | 2 (2.9%) |
| didn't help | 5 (6.9%) | 4 (5.8%) |
| helped only little | 19 (26.4%) | 14 (20.3%) |
| helped | 21 (29.2%) | 22 (31.9%) |
| helped a lot | 22 (30.6%) | 27 (39.1%) |
| Odom | | |
| poor | 11 (14.7%) | 8 (10.8%) |
| fair | 21 (28.0%) | 26 (35.1%) |

| | no recall (N=75) | recall (N=74) |
|--------------------|------------------------|------------------------|
| ood | 33 (44.0%) | 25 (33.8%) |
| xcellent | 10 (13.3%) | 15 (20.3%) |
| )MI improvement | | |
| flean (SD) | 2.289 (2.769) | 3.107 (2.430) |
| fledian (Q1, Q3) | 2.000 (1.000, 5.000) | 3.000 (1.000, 5.000) |
| )I/NDI improvement | | |
| flean (SD) | 13.786 (20.751) | 17.272 (17.953) |
| fledian (Q1, Q3) | 10.500 (1.700, 24.525) | 15.560 (5.800, 29.400) |
| 5D improvement | | |
| flean (SD) | 0.164 (0.403) | 0.200 (0.370) |
| fledian (Q1, Q3) | 0.104 (-0.033, 0.461) | 0.164 (0.000, 0.441) |

```
    Fisher's Exact Test for Count Data
    Kruskal-Wallis rank sum test
    Trend test for ordinal variables
```

```
#(Credits:
#https://rpubs.com/tskam/likert
#https://stackoverflow.com/questions/37761096)

#Making the table long

survey_s <- data %>% filter(!is.na(Satisfaction)) %>%
```

```
group by(group, Satisfaction)%>%summarise(n()) %>%
  pivot wider(names from = Satisfaction, values from = "n()")
survey o <- data %>% filter(!is.na(Outcome)) %>%
  group by(group, Outcome)%>%summarise(n()) %>%
  pivot wider(names from = Outcome, values from = "n()")
survey odom <- data %>% filter(!is.na(Odom)) %>%
 group by(group, Odom)%>%summarise(n()) %>%
  pivot wider(names from = Odom, values from = "n()")
#basic diverging stacked bar chart with percentages as labels
##define a custom panel function (to show and align percentage values)
origNames = colnames(survey s)
myPanelFunc <- function(...) {</pre>
 panel.likert(...)
 vals <- list(...)</pre>
  DF <- data.frame(x=vals$x, y=vals$y, groups=vals$groups)</pre>
  ### some convoluted calculations here...
  grps <- as.character(DF$groups)</pre>
  for(i in 1:length(origNames)){
    grps <- sub(paste0('^',origNames[i]),i,grps)</pre>
  }
  DF <- DF[order(DF$y,grps),]</pre>
  DF$correctX <- ave(DF$x,DF$y,FUN=function(x){</pre>
    x[x < 0] < -rev(cumsum(rev(x[x < 0]))) - x[x < 0]/2
    x[x > 0] \leftarrow cumsum(x[x > 0]) - x[x > 0]/2
    return(x)
  })
```

```
subs <- sub(' Positive$','',DF$groups)</pre>
  \verb|collapse <- subs[-1] == subs[-length(subs)] & DF$y[-1] == DF$y[-length(DF)] \\
$y)]
 DF$abs <- abs(DF$x)</pre>
  DF$abs[c(collapse,FALSE)] <- DF$abs[c(collapse,FALSE)] + DF$abs[c(FALSE,c</pre>
ollapse)]
  DF$correctX[c(collapse, FALSE)] <- 0</pre>
  DF <- DF[c(TRUE,!collapse),]</pre>
  DF$perc <- round(ave(DF$abs,DF$y,FUN=function(x)\{x/sum(x) * 100\}),0)
  panel.text(x=DF$correctX, y=DF$y, label=paste0(DF$perc,'%'), cex=0.7)
}
##stacked bar chart
likert(group ~., survey s, as.percent=TRUE,
       positive.order=FALSE, rightAxis=FALSE,
       main = "Satisfaction",
       xlab="Percentage",
       panel=myPanelFunc)
```

```
origNames = colnames(survey_o)

likert(group ~., survey_o, as.percent=TRUE,
    positive.order=FALSE, rightAxis=FALSE,
    main = "Outcome perceived by the patient",
    xlab="Percentage",
    panel=myPanelFunc,
    auto.key = list(between = 1))
```

```
origNames = colnames(survey_odom)

likert(group ~., survey_odom, as.percent=TRUE,
    positive.order=FALSE, rightAxis=FALSE,
    main = "Outcome perceived by surgeon - Odom criteria",
    xlab="Percentage",
```

```
panel=myPanelFunc,
auto.key = list(between = 1))
```

## Cervical: Patient characteristics by group

- Patients without recall report worse postoperative scores for COMI, ODI/NDI and EQ5D
- Baseline characteristics are similar between the groups
- The outcome of the two groups is similar, as measured by a independent surgeon

| | no recall (N=38) | recall (N=30) |
|--------------------------|-------------------------|-------------------------|
| Gender | | |
| Female | 23 (60.5%) | 20 (66.7%) |
| Male | 15 (39.5%) | 10 (33.3%) |
| Age | | |
| Mean (SD) | 58.579 (9.967) | 58.067 (8.765) |
| Median (Q1, Q3) | 58.000 (49.250, 65.000) | 58.000 (53.000, 63.750) |
| Pathology | | |
| myelopathy | 25 (65.8%) | 20 (66.7%) |
| myelopathy/radiculopathy | 8 (21.1%) | 6 (20.0%) |
| radiculopathy | 5 (13.2%) | 4 (13.3%) |
| ВМІ | | |
| Mean (SD) | 27.233 (3.780) | 27.183 (4.881) |
| Median (Q1, Q3) | 27.320 (25.537, 29.785) | 26.900 (24.770, 28.000) |
| Smoker | | |
| yes | 9 (23.7%) | 6 (20.7%) |
| no | 29 (76.3%) | 23 (79.3%) |
| Segment | | |
| Cervical | 38 (100.0%) | 30 (100.0%) |
| Lumbar | 0 (0.0%) | 0 (0.0%) |
| preop COMI | | |

| | no recall (N=38) | recall (N=30) |
|-----------------|-------------------------|-------------------------|
| Mean (SD) | 7.368 (2.174) | 6.893 (2.039) |
| Median (Q1, Q3) | 8.000 (6.000, 9.000) | 7.000 (6.000, 8.000) |
| preop ODI/NDI | | |
| Mean (SD) | 47.639 (18.639) | 41.914 (17.581) |
| Median (Q1, Q3) | 54.000 (31.325, 63.550) | 44.000 (32.000, 55.000) |
| preop EQ5D | | |
| Mean (SD) | 0.385 (0.328) | 0.523 (0.239) |
| Median (Q1, Q3) | 0.516 (0.010, 0.612) | 0.586 (0.516, 0.689) |
| postop COMI | | |
| Mean (SD) | 5.622 (2.639) | 3.704 (2.267) |
| Median (Q1, Q3) | 5.000 (4.000, 8.000) | 4.000 (2.000, 5.000) |
| postop ODI/NDI | | |
| Mean (SD) | 40.422 (18.763) | 24.500 (16.962) |
| Median (Q1, Q3) | 42.000 (28.000, 54.000) | 25.200 (11.500, 36.150) |
| postop EQ5D | | |
| Mean (SD) | 0.494 (0.301) | 0.661 (0.273) |
| Median (Q1, Q3) | 0.516 (0.452, 0.691) | 0.689 (0.585, 0.837) |
| ucation | | |

| | no recall (N=38) | recall (N=30) |
|---|---|---|
| <=4 | 14 (50.0%) | 6 (28.6%) |
| >4 | 14 (50.0%) | 15 (71.4%) |
| Satisfaction.numeric | | |
| Mean (SD) | 4.649 (0.824) | 4.852 (0.362) |
| Median (Q1, Q3) | 5.000 (5.000, 5.000) | 5.000 (5.000, 5.000) |
| Outcome.numeric | | |
| Mean (SD) | 3.568 (1.119) | 4.111 (0.751) |
| Median (Q1, Q3) | 4.000 (3.000, 4.000) | 4.000 (4.000, 5.000) |
| Odom.numeric | | |
| Mean (SD) | 2.500 (0.797) | 2.567 (0.817) |
| Median (Q1, Q3) | 3.000 (2.000, 3.000) | 2.500 (2.000, 3.000) |
| Satisfaction | | |
| N-Miss | 1 | 3 |
| very dissatisfied | 1 (2.7%) | 0 (0.0%) |
| somewhat dissatisfied | 0 (0.0%) | 0 (0.0%) |
| neither satisfied or dissatisfied | 2 (5.4%) | 0 (0.0%) |
| somewhat satisfied | 5 (13.5%) | 4 (14.8%) |
| very satisfied | 29 (78.4%) | 23 (85.2%) |

| | no recall (N=38) | recall (N=30) |
|---------------------|------------------------|------------------------|
| Outcome | | |
| N-Miss | 1 | 3 |
| made things worse | 2 (5.4%) | 0 (0.0%) |
| didn't help | 3 (8.1%) | 0 (0.0%) |
| helped only little | 13 (35.1%) | 6 (22.2%) |
| helped | 10 (27.0%) | 12 (44.4%) |
| helped a lot | 9 (24.3%) | 9 (33.3%) |
| Odom | | |
| poor | 5 (13.2%) | 2 (6.7%) |
| fair | 11 (28.9%) | 13 (43.3%) |
| good | 20 (52.6%) | 11 (36.7%) |
| excellent | 2 (5.3%) | 4 (13.3%) |
| COMI improvement | | |
| Mean (SD) | 1.865 (2.771) | 3.141 (2.125) |
| Median (Q1, Q3) | 2.000 (0.000, 5.000) | 3.000 (1.500, 4.500) |
| ODI/NDI improvement | | |
| Mean (SD) | 6.992 (15.900) | 16.375 (17.515) |
| Median (Q1, Q3) | 5.600 (-4.000, 20.000) | 14.500 (5.900, 28.925) |

### **EQ5D** improvement

Mean (SD) 0.106 (0.383) 0.138 (0.302)

Median (Q1, Q3) 0.070 (-0.044, 0.436) 0.104 (0.000, 0.272)

summary(tab 2, pfootnote=TRUE)

```
1. Fisher's Exact Test for Count Data
```

- 2. Kruskal-Wallis rank sum test
- 3. Trend test for ordinal variables

```
#compare means of satisfaction and outcomes questions of postoperative COMI
(as numeric)
plot6a <- cervical %>% ggplot(aes(group, Outcome.numeric)) +
                   geom boxplot(width=0.2, fill = "#1f78b4", alpha=0.8) +
                   stat compare means(label.x=1) +
                   theme bw()
plot6b <- cervical %>% ggplot(aes(group, Satisfaction.numeric)) +
                   geom boxplot(width=0.2, fill = "#1f78b4", alpha=0.8) +
                   stat_compare_means(label.x=1) +
                   theme_bw()
plot6c <- cervical %>% ggplot(aes(group, Odom.numeric)) +
                   geom boxplot(width=0.2, fill = \#1f78b4, alpha=0.8)+
                   stat compare means(label.x=1) +
                   theme bw()
plot6 <- plot6a + plot6b + plot6c + plot_annotation(tag_levels = 'A')</pre>
plot6
```

```
#Making the table long
csurvey s <- cervical %>% filter(!is.na(Satisfaction)) %>%
 group by (group, Satisfaction) %>%summarise(n()) %>%
  pivot wider(names from = Satisfaction, values from = "n()")
csurvey o <- cervical %>% filter(!is.na(Outcome)) %>%
 group by(group, Outcome)%>%summarise(n()) %>%
 pivot wider(names from = Outcome, values from = "n()")
csurvey odom <- cervical %>% filter(!is.na(Odom)) %>%
 group by(group, Odom)%>%summarise(n()) %>%
  pivot_wider(names_from = Odom, values_from = "n()")
#input values to solve NA problem
csurvey s[2,2] <- 0
csurvey s[2,3] < 0
csurvey o$`made things worse` <- as.double(csurvey o$`made things worse`)</pre>
csurvey_o$`didn't help` <- as.double(csurvey_o$`didn't help`)</pre>
csurvey o[2,2] <- 0.0001
csurvey o[2,3] < -0.0001
#basic diverging stacked bar chart with percentages as labels
origNames = colnames(csurvey s)
```

```
likert(group ~., csurvey_s, as.percent=TRUE,
    positive.order=FALSE, rightAxis=FALSE,
    main = "Satisfaction",
    xlab="Percentage",
    panel=myPanelFunc)
```

#### Satisfaction



```
origNames = colnames(csurvey_o)

likert(group ~., csurvey_o, as.percent=TRUE,
    positive.order=FALSE, rightAxis=FALSE,
    main = "Outcome perceived by the patient",
    xlab="Percentage",
    panel=myPanelFunc,
    auto.key = list(between = 1))
```

### Outcome perceived by the patient



```
origNames = colnames(csurvey_odom)

likert(group ~., csurvey_odom, as.percent=TRUE,
    positive.order=FALSE, rightAxis=FALSE,
    main = "Outcome perceived by surgeon - Odom criteria",
    xlab="Percentage",
    panel=myPanelFunc,
    auto.key = list(between = 1))
```

### Outcome perceived by surgeon - Odom criteria

